CLINICAL TRIAL: NCT00549211
Title: A Two-Part Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Repeat Oral Doses of GSK557296 in a Randomized, Single-Blind, Placebo-Controlled, Dose-Rising Design, and to Evaluate the Effect of Food on Single Oral Doses of GSK557296 in Healthy Adult Subjects
Brief Title: A First Time in Human Study in Healthy Male Volunteers for Compound GSK557296.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OTB109039
Record Dates: First submitted 2007-10-23; First posted 2007-10-25 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Obstetric Labour, Premature; Premature Ejaculation
Keywords: Healthy Subjects,; Safety,; Tolerability,; Pharmacokinetics
MeSH Terms: conditions — Premature Birth; Premature Ejaculation | interventions — epelsiban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK557296

SUMMARY:
A study conducted on healthy volunteers to determine the safety, tolerability and affect on the human body by experimental drug GSK557296.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males who are 18 to 45 years of age
* Body mass index between 19 and 30 with a body weight greater than 110 pounds and deemed healthy by a physician
* Non-smokers

Exclusion Criteria:

* Alcohol consumption averaging more than 7 drinks per week
* Positive for Hepatitis C antibody, Hepatitis B antigen or HIV
* Any use of prescription drugs or non prescription drugs

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2007-10

PRIMARY OUTCOMES:
Safety tests up to 24 hrs after dose 12-lead ECG to look at the heart prior to dose and up to 24 hours after Dual-lead telemetry to monitor the heart rhythms for 20 hours prior to dosing and up to 12 hours after dosing Periodic vital signs | 24 Hours

SECONDARY OUTCOMES:
Blood tests to study how long the drug stays in your blood | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Evansville, Indiana, United States